CLINICAL TRIAL: NCT00589264
Title: Zinc and Biobehavioral Development in Early Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Instituto de Investigacion Nutricional, Peru (Other); University of Kansas (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Laura Caulfield, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5R01HD045430 (NIH); 5R01HD045430 (NIH)
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Child Development
Keywords: zinc; iron; child development; visual attention; Peru
MeSH Terms: interventions — Zinc; Iron; Copper

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): iron + copper + zinc
  Interventions: Dietary Supplement: zinc
- 2 (Active Comparator): iron + copper only
  Interventions: Dietary Supplement: iron + copper

INTERVENTIONS:
Dietary Supplement: zinc — 10 mg elemental zinc + 10 mg elemental iron + 0.5 mg copper syrup taken daily for 1 year, from 6 to 18 months of age
  Arms: 1
Dietary Supplement: iron + copper — 10 mg elemental iron + 0.5 mg copper in syrup given daily for one year from 6 months to 18 months of age
  Arms: 2

SUMMARY:
Zinc is necessary for growth and development, including the central nervous system, and zinc deficiency which is common in resource-poor settings, may adversely affect social, behavorial, cognitive and sensorimotor development. The project, located in Lima Peru, utilizes an experimental model in which children receive 10 mg supplemental zinc (or not) daily along with 10 mg iron and 1/2 mg copper from 6 months of age to 18 months of age. Beginning at 6 months of age, and at 9, 12, and 18 months, children are evaluated in multiples aspects of development. Children are also followed for their diet, growth, and health status. We hypothesize that children in this setting in which the diet is low in zinc who receive supplemental zinc will have better information processing skills, sensorimotor and behavioral development than their counterparts who do not receive supplemental zinc.

ELIGIBILITY:
Inclusion Criteria:

* Born at term of non-low birth weight
* Free of major malformations, genetic abnormalities or health problems associated with developmental delays
* Planning to remain in study area for one year
* In good general health

Exclusion Criteria:

* Low birth weight
* Non-term delivery
* Vision or hearing problems
* Anemia

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
cognitive development(visual attention, executive processing, vigilance) | 6, 9, 12, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Caulfield, PhD, Principal Investigator — Johns Hopkins Bloomberg SPH
Locations (1):
- Instituto de Investigacion Nutricional, Lima, Peru

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923
- [Derived] Colombo J, Zavaleta N, Kannass KN, Lazarte F, Albornoz C, Kapa LL, Caulfield LE. Zinc supplementation sustained normative neurodevelopment in a randomized, controlled trial of Peruvian infants aged 6-18 months. J Nutr. 2014 Aug;144(8):1298-305. doi: 10.3945/jn.113.189365. Epub 2014 May 21. PMID 24850625